CLINICAL TRIAL: NCT00027339
Title: A Phase II Study of the Predictive Value of Pharmacokinetic-Adjusted Phenotypic Susceptibility (C12h/IC50) on Antiretroviral Response to Ritonavir-Enhanced Protease Inhibitors in Subjects With Failure of Previous Protease Inhibitor-Based Regimens
Brief Title: Using Drug Levels and Drug Resistance Testing to Select Effective Anti-HIV Drug Combinations in Patients With Drug-resistant HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5126; 10079 (Registry Identifier: DAIDS ES); ACTG A5126; AACTG A5126
Record Dates: First submitted 2001-12-04; First posted 2001-12-05 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV-1; HIV Protease Inhibitors; RNA, Viral; Phenotype; Viral Load; Pharmacokinetics; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Indinavir; Tenofovir; Ritonavir; fosamprenavir

INTERVENTIONS:
Drug: lopinavir/ritonavir
Drug: indinavir sulfate
Drug: tenofovir disoproxil fumarate
Drug: ritonavir
Drug: fosamprenavir

SUMMARY:
Because people infected with HIV strains that are resistant to anti-HIV drugs have fewer effective treatment options, selecting an effective anti-HIV drug combination is difficult. A combination of protease inhibitors (PIs), when added to a patient's current anti-HIV therapy, may decrease viral load and increase drug activity. Tests that measure drug levels in the blood and tests to evaluate the drug resistance of HIV may also be helpful in choosing the best anti-HIV drug combination for a patient. This study will determine whether using these tests to choose a drug combination and adding PIs to that combination will improve the patient's response to anti-HIV therapy.

DETAILED DESCRIPTION:
Treatment options are limited for HIV infected individuals who have extensive treatment experience and harbor resistance to antiretrovirals (ARVs) from multiple drug classes. Increasing the concentration of PIs in a regimen may be one way to provide more substantial ARV activity. It is uncertain how combining specific PIs with RTV affects viral susceptibility and ARV effect. The relationship of PI concentration (e.g., Cmin) to virus susceptibility (IC50) may be a better predictor of treatment outcome than susceptibility alone. This study will evaluate the predictive value of pharmacokinetic-adjusted phenotypic susceptibility (C12h/IC50) on ARV response to ritonavir (RTV)-boosted regimens in patients failing their current PI-containing regimens.

Participants will have blood drawn during a screening visit for phenotypic assay and to determine viral load. At study entry, participants will discontinue their PIs while continuing to take their other ARVs. Each participant and his or her doctor will choose to add one of three RTV-boosted regimens: 1) indinavir (IDV) and RTV; 2) fosamprenavir (FPV) and RTV; or 3) lopinavir (LPV)/RTV plus additional RTV. Participants will take this regimen for 14 days. On Day 14, patients will have a 12-hour pharmacokinetic evaluation. On Day 15, patients will add tenofovir disoproxil fumarate (TDF) to their regimens and may choose to modify their other ARVs while continuing their RTV-boosted therapy. Participants will have additional study visits at Weeks 4, 8, 16, and 24. Study visits will include a physical exam and blood and urine tests. Participants will complete adherence questionnaires four times during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Viral load greater than 2500 copies/ml within 60 days of study entry
* On regimen with at least one PI for a total of at least 48 weeks
* On the same PI regimen for at least 90 days prior to study entry
* Decreased susceptibility to two of these three PIs: LPV, APV, and IDV (documented by phenotype within 90 days prior to study entry)
* Have taken a nonnucleoside reverse transcriptase inhibitor (NNRTI) for at least 12 weeks anytime in previous treatment history, or have decreased susceptibility to at least two NNRTIs
* Have taken two or more nucleoside reverse transcriptase inhibitors (NRTIs) for at least 12 weeks anytime in previous treatment history
* Agrees to use acceptable methods of contraception
* Weighs 88 lbs or more

Exclusion Criteria:

* Cannot tolerate RTV, APV, FPV, LPV/RTV, or IDV
* Use of HIV vaccines, investigational agents, hydroxyurea, or therapy to affect the immune system within 60 days of study entry
* Serious kidney problems
* Pregnancy or breastfeeding
* Alcohol or drug use that would interfere with the study
* Serious illness that requires treatment or hospitalization (patients stable on therapy or who have finished therapy at least 14 days before study entry may be eligible)

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Richman, MD, Study Chair — University of California, San Diego; Joseph J. Eron, MD, Study Chair — University of North Carolina, Chapel Hill
Locations (14):
- United States (13):
  - USC CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - Ucsd, Avrc Crs, San Diego, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico